CLINICAL TRIAL: NCT02437500
Title: Expanded Access Program of SER-109 in the Treatment of Adults With Recurrent Clostridioides Difficile Infection (RCDI)
Status: Approved for marketing | Type: Expanded Access
Sponsor: Seres Therapeutics, Inc. (Industry)
Responsible Party: Sponsor
Other Study IDs: SERES-016
Record Dates: First submitted 2015-05-05; First posted 2015-05-07 (Estimated); Last update posted 2023-06-13 (Actual); Status verified 2023-06

CONDITIONS: Clostridioides Difficile Infection
Keywords: Clostridioides Difficile Infection; Gastrointestinal Diseases; Digestive System Diseases; Intestinal Diseases; Gram-Positive Bacterial Infections; Communicable Diseases
MeSH Terms: conditions — Clostridium Infections; Gastrointestinal Diseases; Digestive System Diseases; Intestinal Diseases; Gram-Positive Bacterial Infections; Communicable Diseases

STUDY DESIGN:
Expanded Access Types: Treatment

INTERVENTIONS:
Biological: SER-109 — SER-109 is an ecology of bacteria in spore form, enriched from stool donations obtained from healthy, screened donors
  Other Names: Eubacterial Spores, Purified Suspension, Encapsulated

SUMMARY:
Subjects will receive an oral dose of SER-109 in 4 capsules once daily for 3 consecutive days. The purpose of this study is to provide access to SER-109 for adult subjects with recurrent Clostridioides Difficile Infection (RCDI) and to monitor subject safety and report to regulatory authorities, as appropriate.

DETAILED DESCRIPTION:
SERES-016 is a multicenter, expanded-access program (EAP) of SER-109 for subjects with RCDI conducted in the US. Up to approximately 90 subjects are expected to be treated with SER-109, or until SER-109 investigational product is exhausted. Within 3 days after end of antibiotics and on the day preceding SER-109, a bowel cleanse should be administered.

Subjects who meet all the inclusion criteria and none of the exclusion criteria are eligible for participation in the EAP. Each subject (or subject's legally authorized representative) will have to sign an informed consent form (ICF) indicating their consent to participate in the EAP.

Subjects will receive an oral dose of SER-109 in 4 capsules once daily for 3 consecutive days.

ELIGIBILITY:
Main Inclusion Criteria:

1. Signed informed consent prior to initiation of any EAP-specific procedure or treatment. The subject, or their legally authorized representative, must be willing to provide written informed consent and understand the potential risks and benefits from EAP enrollment and treatment.
2. ≥2 episodes of CDI inclusive of the current episode
3. The CDI recurrence must have met the protocol definition of:

   1. ≥3 unformed stools per day for 2 consecutive days
   2. A positive C. difficile stool toxin assay or PCR test
   3. CDI antibiotic therapy defined as either 10-21 days of vancomycin (125 mg po QID) or fidaxomicin (200 mg po BID). Pulse taper courses are also accepted.
   4. An adequate clinical response to antibiotic therapy, defined as (<3 unformed stools in 24 hours) for 2 or more consecutive days while on antibiotics.
   5. The requirement that the subject can be dosed with study drug within 4 days of antibiotic completion.

Main Exclusion Criteria:

1. Female subjects who are pregnant, breastfeeding, lactating, or planning to become pregnant during the study.
2. Known or suspected toxic megacolon and/or known small bowel ileus.
3. Admitted to or expected to be admitted to an intensive care unit.
4. Absolute neutrophil count of <500 cells/mm^3.
5. Major gastrointestinal surgery (e.g., significant bowel resection or diversion) within 3 months before enrollment (this does not include appendectomy or cholecystectomy), or any history of total colectomy or bariatric surgery (bariatric surgery which does not disrupt the gastrointestinal lumen, i.e., restrictive procedures such as banding, are permitted).
6. History of active inflammatory bowel disease (ulcerative colitis, Crohn's disease, microscopic colitis) with diarrhea believed to be caused by active inflammatory bowel disease in the past 3 months.
7. Any history of fecal microbiota transplantation (FMT) in the past 3 months.
8. Concurrent intensive induction chemotherapy, radiotherapy, or biologic treatment for active malignancy (subjects on maintenance chemotherapy may only be enrolled after consultation with the study medical monitor).

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult